CLINICAL TRIAL: NCT03050957
Title: Effect of Oral Menthol on the Swallow Response of Patients With Oropharyngeal Dysphagia Associated With Neurological Diseases and Aging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, PhD, MD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA01-11//2012
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- menthol 10 mM (millimolar) (Experimental): Patients were studied during the deglutition of one series of 5, 10 and 20 mL nectar control boluses and two series of 5, 10 and 20 mL nectar boluses supplemented with the corresponding concentration of menthol 10 mM
  Interventions: Dietary Supplement: menthol
- menthol 1 mM (Experimental): Patients were studied during the deglutition of one series of 5, 10 and 20 mL nectar control boluses and two series of 5, 10 and 20 mL nectar boluses supplemented with the corresponding concentration of menthol 1 mM
  Interventions: Dietary Supplement: menthol

INTERVENTIONS:
Dietary Supplement: menthol — Alimentary bolus supplemented with menthol

SUMMARY:
Oropharyngeal dysphagia (OD) is the most frequent digestive disorder in older people (>70 years) and has been recently recognized as a geriatric syndrome. The main features of OD are: a high prevalence and severe complications either related with the decreased swallowing efficacy with 45% prevalence of malnutrition or due to decreased swallowing safety with 50% prevalence of aspiration pneumonia that increases hospital stay by 100% and leads to a 50% of mortality rate. However, there is no specific pharmacologic treatment for OD in older patients yet. Treatments are now evolving from compensation to active treatments aiming to restore the swallowing dysfunction and some groups have been looking for new therapeutic strategies. The main goal of this study is to evaluate the effect of administering menthol in bolus on the swallowing response in elderly and neurogenic patients with OD. In addition, this study will also assess the side effects of this pharmacological strategy.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspicion of OD associated with aging (>70 years), neurodegenerative diseases or stroke.

Exclusion Criteria:

* Patients with suspicion that they will not be able to compliment the protocol, patients participating or have participated in a clinical study the last 4 weeks and patients with alcoholic or drugs dependence

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Laryngeal vestibule closure time | Laryngeal vestibule closure time is assessed during the videofluoroscopic assessment. Laryngeal vestibule closure time can occur between 100 milliseconds from the GPJ opening up to 1000 milliseconds.
  timing of the opening of the laryngeal vestibule (LV), glossopalatine junction (GPJ) opening being given the time value 0

IPD SHARING:
Plan to Share IPD: No